CLINICAL TRIAL: NCT05762575
Title: Application of New Knotting Methods in Single-hole Laparoscopic Suturing Instructional Program on the Basis of Multidirectional Stitching Technology
Brief Title: Application of Spaghetti Knotting Technology in Single-hole Laparoscopic Suturing Instructional Program on the Basis of Multidirectional Stitching Technology.
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2022-07-205
Record Dates: First submitted 2023-02-23; First posted 2023-03-09 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Knotting Methods; Single-port Laparoscopic Surgery

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: The volunteers in control group study traditional knotting technology,
  Interventions: Other: knotting methods
- new knotting group: The volunteers in experimental group study new knotting technology.
  Interventions: Other: knotting methods

INTERVENTIONS:
Other: knotting methods — The volunteers in experimental group study new knotting technology.

SUMMARY:
The surgeon's knot-tying technique plays a crucial role in the recovery of patients after single-port laparoscopy. Knot tying is very challenging in minimally invasive surgery and is a critical skill in advanced surgery. In this study, investigators introduce a new knotting technique, compare it with the traditional knotting technique in many aspects, and also discuss its application in the teaching of single-port laparoscopic knotting.

ELIGIBILITY:
Inclusion Criteria:

1. the habitual hand is the right hand;
2. no practical experience in operating single-hole laparoscopic instruments;
3. no simulator sickness;
4. training and assessment are completed on time and carefully

Exclusion Criteria:

1. have participated in other skills training programs
2. are not interested in single-hole laparoscopy will be excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the candidates were junior residents. Forty volunteers were selected according to the established criteria and randomly divided into control group and experimental group by computer-generated simple randomization. There were twenty volunteers in each group, and each group was composed of five males and fifteen females. The volunteers in control group study traditional knotting technology, and the volunteers in experimental group study new knotting technology. A statistician in our hospital completed the random distribution of the subjects and ensured the confidentiality of the grouping information. Before participating in the study, the subjects completed a questionnaire about their demographic information, such as age, gender and experience in video games.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Accuracy of needle entry | through study completion, an average of 1 month
  The needle stick should be in and out of the centre of the dot. The operator received 2 points if it was in the centre of the dot, 1 point if it deviated from the centre, and 0 points if it was outside the dot.
Stability of the knot | through study completion, an average of 1 month
  The knot was required to be a surgical triple knot and should not have been a smooth knot or a loose knot. A normal knot received 2 points. A smooth knot received 1 point,and 0 points were awarded for a loose knot.
Tissue integrity | through study completion, an average of 1 month
  The suture tissue should not be damaged or ruptured. The trainee received a score of two for integrity, 1 for a few cracks, and 0 for a complete fracture of the tissue.
Tightness of the tissue | through study completion, an average of 1 month
  The tightness of the suture tissue indicated that the two sides of the sutured tissue were closely connected. The operator received 2 points if there was no gap between the two sides of the incision, 1 point for a few gaps, and 0 points for a totally loose suture.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Zhejiang, China